CLINICAL TRIAL: NCT04999787
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial Evaluating the Efficacy, Safety, and Pharmacokinetics of HSK21542 Injection in Liver Disease Subjects With Pruritus
Brief Title: A Clinical Trial Evaluating the Efficacy, Safety, and Pharmacokinetics of HSK21542 Injection in Liver Disease Subjects With Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK21542-204
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK21542 (Experimental): HSK21542-0.3 μg/kg，HSK21542-0.6 μg/kg
  Interventions: Drug: HSK21542
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK21542 — HSK21542-0.3 μg/kg，HSK21542-0.6 μg/kg
  Arms: HSK21542
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a multi-center, randomized, double-blind, placebo-controlled study. About 90 liver disease subjects with moderate or above pruritus are planned to be enrolled. They will be randomized to two dose groups (0.3 μg/kg and 0.6 μg/kg) and a placebo control group at a 1:1:1 ratio, with about 30 subjects in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 and ≤ 75 years old, male or female;
2. Body mass index (BMI): ≥ 18 kg/m2 and ≤ 35 kg/m2;
3. Suffering from liver diseases with itching, including but not limited to viral hepatitis, autoimmune liver disease, drug-induced liver disease, alcoholic liver disease, and other liver diseases;
4. The mean baseline WI-NRS score before randomization suggests moderate to severe itching (≥ 4 points) and the last two WI-NRS scores ≥ 4 points.
5. Subjects who are willing to sign an informed consent form in written form fully understand the objectives and purposes of the study, and are willing to comply with the study protocol before any of the study-related procedures to start.

Exclusion Criteria:

1. Decompensated hepatic cirrhosis in the following cases:

   1. History of liver transplant, expecting a liver transplant surgery, or the current model for end-stage liver disease (MELD) score ≥ 18;
   2. Grade 3 ascites;
   3. History of gastrointestinal hemorrhage (excluding haemorrhoidal haemorrhage) within one month before randomization;
   4. Hepatic encephalopathy;
2. Having dermatitis atopic, chronic urticaria, psoriasis or other skin diseases that the investigator determines will disturb the assessment of itching or having itching caused by other diseases.
3. History of allergy to opioids, such as urticaria;
4. Cannot ensure the stable use of drugs for the treatment of baseline liver diseases from 4 weeks before the lead-in phase to the end of the follow-up period, such as ursodeoxycholic acid (UCDA), antiviral drugs (excluding interferon), fibrates, etc.;
5. Cannot ensure the stable use of drugs that may affect the efficacy or safety evaluations from the first 14 days of the lead-in phase to the end of the follow-up period, such as antipsychotics, sedative hypnotics, anxiolytics, antidepressants (excluding selective serotonin reuptake inhibitors), immunosuppressants/immunomodulators (such as systemic glucocorticoid therapy [excluding topical application], ciclosporin A, azathioprine, methotrexate, etc.);
6. Using drugs with unclear half-life that may affect the efficacy evaluation within 14 days before the lead-in period, or drugs that affect the efficacy evaluation before randomization, and the last time of use is shorter than 5 half-lives from the lead-in phase (refer to the specific drug labeling), including but not limited to bile acid binding resin (colestyramine, etc.), pregnane X receptor (PXR) agonist (rifampicin, etc.), selective serotonin reuptake inhibitor (SSRIs) (sertraline, etc.), antihistamines, gabapentin, pregabalin, interferon, obeticholic acid or other opioids;
7. Using the following topical drugs within 3 days before the lead-in phase: antihistamines and glucocorticoids;
8. Having received traditional Chinese medicine treatment, physical phototherapy or artificial liver treatment that may affect the efficacy evaluation within 14 days before randomization;
9. Complicated with other serious underlying diseases that the investigator judges may increase the risk of the trial, affect the compliance of the subjects with the protocol or affect the subjects with completion of the trial, including but not limited to malignant tumors (excluding tumors that had been cured [no evidence of disease recurrence within 5 years]), serious cardiovascular and cerebrovascular diseases, mental and neurological disorders, etc.;
10. Complicated with uncontrolled severe infections (including severe abdominal infection, upper respiratory tract infection, lower respiratory tract infection, urinary system infection, etc.);
11. Itching secondary to obstruction of bile duct (excluding primary sclerosing cholangitis (PSC));
12. With the following abnormal laboratory tests results:

    1. eGFR < 30 mL/min/1.73 m2;
    2. Serum bilirubin total (TBIL) > 15 × ULN;
    3. INR > 1.5 × ULN;
    4. Potassium ion concentration < 3.0 mmol/L;
13. History of medication or drug abuse and/or alcohol abuse within 3 months prior to screening (alcohol abuse is defined as an average of > 2 units of alcohol consumed per day [1 unit = 360 mL of beer with 5% alcohol, 45 mL of liquor with 40% alcohol, or 150 mL of wine] within 3 months);
14. Having participated in other clinical trials within 3 months prior to screening (defined as having received investigational drug or placebo);
15. Positive for human immunodeficiency virus (HIV) antibody or syphilis antibody at screening;
16. Pregnant and breastfeeding females; women of child-bearing potential or men who are unwilling to use contraception during the trial; or subjects who are planning pregnancy within 3 months after the completion of the trial (including male subjects);
17. Expected survival < 3 months;
18. Subjects judged by the investigator to have any other factors unsuitable for involvement in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Changes in daily Worst Itching Intensity Numerical Rating Scale (WI-NRS) scores from baseline during the administration period | Day 1 to Day 28
  In the NRS score, 0-10 represents different degrees of itching, the larger the number, the more severe the itching
The proportion of subjects whose daily WI-NRS scores improve by ≥ 3 points and ≥ 4 points compared with baseline during the administration period | Day 1 to Day28
Area under curve (AUC) of daily WI-NRS scores during the administration period | Day 1 to Day28
Changes in WI-NRS per unit time (per day) from baseline during the administration period | Day 1 to Day 28
Changes in quality of life (evaluated by Skindex-16 scale) from baseline during the administration period | Day 1 to Day 28
Changes in daily WI-NRS scores from baseline during the follow-up period | Day 29 to Day 31

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, China